CLINICAL TRIAL: NCT01647425
Title: Prevalence and Risk Factors for Persistent Tobacco or Alcohol Use Over the First Year of a First Lung or Head and Neck Cancer
Brief Title: Alcohol and Tobacco Consumption in Patients With Head and Neck or Lung Cancer
Acronym: ALTAK
Status: Completed | Type: Observational
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Centre Régional de Référence en Cancérologie (Other); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: ALTAK - 1109
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2014-08

CONDITIONS: Head and Neck Cancer; Lung Cancer
Keywords: head and neck cancer; lung cancer; tobacco use disorder; alcoholism
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Tobacco Use Disorder; Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- head and neck or lung cancer: patient with a first head and neck cancer or first lung cancer
  Interventions: Behavioral: physician assessment

INTERVENTIONS:
Behavioral: physician assessment — * Socio-economic conditions and general features: educational level, professional status...
  * Assessment of current and past use of tobacco: current smoking status reported by the patient; in lifelong non-smokers: previous history of passive smoking reported by the patient; breath carbon monoxide level; in past smokers: age of first cigarette, total reported duration of active smoking, breath carbon monoxide level...
  * in current smokers: age of first tobacco use, total reported duration of active smoking; Fagerström Nicotine Dependence Test...
  * Assessment of the current and past uses of alcohol: previous-year assessment using the CAGE questionnaire and the AUDIT Test; average weekly alcohol consumption over the last 12 months...
  * Assessment of current use of cannabis using the Cannabis Abuse Screening Test
  * Psychiatric assessment using the MINI 5.0

SUMMARY:
This is an multicenter study for preventive and therapeutic strategies for patients with head and neck cancer

DETAILED DESCRIPTION:
Continuing the chronic intoxication by either tobacco or alcohol after the initial diagnosis of a first lung or head and neck cancer significantly improves the risk of experiencing a second cancer, and largely affects the long term survival. Addiction intervention programs should be personalized according to the patient's profile, with the aim to develop more sustained intervention and monitoring in patients identified at higher risk of not spontaneously stopping harmful substance use. As of today, the trajectories of smoking and drinking habits and the risk factors for persisting smoking or drinking habits have been insufficiently explored among patients with a first lung or head and neck cancer.

The ALTAK study aims to depict the rate of tobacco smokers 12 months after the initial diagnosis of a first lung or head and neck cancer. The secondary objectives of the study are:

* to depict the rate of alcohol users 12 months after the initial diagnosis of a H&N cancer
* to depict the rate of tobacco smokers at cancer diagnosis
* to depict the rate of alcohol users at cancer diagnosis
* to determine the social, motivational, psychiatric, tobacco-related, alcohol-related, and cannabis-related features associated with stopping tobacco in the year following the diagnosis of a first TARC.
* to determine the social, psychiatric, tobacco-related, alcohol-related, and cannabis-related features associated with stopping alcohol drinking in the year following the diagnosis of a first H&N cancer

ELIGIBILITY:
Inclusion Criteria:

* first head and neck or lung cancer
* first support
* age ≥ 18
* patient covered by health insurance
* signed informed consent

Exclusion Criteria:

* prior lung or head and neck cancer
* History of another cancer <5 years, not evolutive and untreated at baseline (carcinoma of the cervix, or basal cell carcinoma of the skin properly treated are allowed). The presence of a second discovery tumor location at the same time as the lung or head and neck cancer, is not a criteria for non-inclusion
* mesothelioma and oesophageal cancer
* unable to undergo trail medical follow up (geographical, social and psychological reasons)
* pregnant or nursing women
* patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with a first head and neck cancer or first lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
tobacco consumption | at 12 months
  reported tobacco smoking

SECONDARY OUTCOMES:
tobacco smoking | at baseline, 3 and 6 months
  frequency tobacco consumption
alcohol drinking | at baseline, 3, 6 and 12 months
  frequency of alcohol consumption
progression free survival | at 12 months
  median time between date of inclusion and date of first progression
overall survival | at 12 months
  median time between date of inclusion and date of death
sociodemographic, cancer-related, tobacco-related, alcohol-related, and psychiatric characteristics | at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Corinne VANNIMENUS, MD, Study Director — Centre Hospitalier Régional et Universitaire LILLE
Locations (3):
- France (3):
  - Centre Hospitalier Régional et Universitaire - Hopital CALMETTE, Lille
  - Centre Hospitalier Régional et Universitaire - Hopital HURIEZ, Lille
  - Oscar Lambret Center, Lille

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vannimenus C, Bricout H, Le Rouzic O, Mouawad F, Chevalier D, Dansin E, Rotsaert L, Lefebvre G, Cottencin O, Porte H, Scherpereel A, El Fahsi A, Richard F, Rolland B; ALTAK Study Group. Compared characteristics of current vs. past smokers at the time of diagnosis of a first-time lung or head and neck cancer: a cross-sectional study. BMC Cancer. 2018 Apr 3;18(1):372. doi: 10.1186/s12885-018-4253-5. PMID 29614983